CLINICAL TRIAL: NCT04423835
Title: Applying Paley's Principles to Lateral Closing Wedge Osteotomy for Cubitus Varus Deformity in Children
Brief Title: Lateral Closing Wedge Osteotomy for Cubitus Varus Deformity in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuxi Su, Vice professor, Children's Hospital of Chongqing Medical University
Other Study IDs: CQMU20200026
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Deformity; Bone
Keywords: cubitus varus; supracondylar humerus fracture; osteotomy
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lateral closing osteotomy for cubitus varus deformity: The osteotomy line of all patients was designed according to Paley's principles. The lateral incision was applied in all patients and the osteotomy lines were marked on the humerus with the assistance of C-arm radiographs.
  Interventions: Procedure: Paley's Principle osteotomy

INTERVENTIONS:
Procedure: Paley's Principle osteotomy — . The osteotomy line of all patients was designed according to Paley's principles. The lateral incision was applied in all patients and the osteotomy lines were marked on the humerus with the assistance of C-arm radiographs. An isosceles triangle template was used for osteotomy, and the medial cortex was left intact. K-wires were used to fix the osteotomy laterally.
  Other Names: Applying Paley's Principles to Lateral Closing Wedge Osteotomy

SUMMARY:
Humeral osteotomy is the most effective method for evident cubitus varus correction in children. Several osteotomy methods and fixation materials have been developed in the past. By applying the principles of deformity correction described by Paley, the investigators describe a novel corrective technique for cubitus varus involving lateral osteotomy using Kirschner wires.

DETAILED DESCRIPTION:
Supracondylar humerus fractures (SHFs) account for approximately 10% of all pediatric fractures in children. Poorly treated SHFs can lead to the most common cubitus varus deformity especially in patients treated conservatively. The cosmetic aspect of this deformity is the main concern of patients, together with reduced remodeling ability. Inevitably, surgery is the first choice for such patients. Several osteotomy techniques and fixation materials have been developed in the last several decades. With the advent of three-dimensional printing techniques and computed tomography reconstruction methods, more accurate computing designs have been applied in the correction of cubitus varus. These techniques make the surgery more complex and require the performance of computed tomography (CT), resulting in high radiation exposure in children. Paley described the principles of deformity correction that are widely used for the lower limbs. These principles represent an alternative with easy application without the need of CT, with less occurrence of prominence and good cosmetic outcome. According to the Paley principles, all the vertex of the triangular osteotomy should site on the center of rotation of angulation (CORA) line, by doing this, the gun-butt deformity was corrected perfectly. More importantly, they help to accurately correct the anatomic axis of the upper limb. According to our knowledge, this is the first study describes the lateral closing wedge osteotomy for correction cubitus varus deformity in children by applying Paley's principles and fixation with K-wires.

Taken together, the investigators aimed at verifying the feasibility of Paley's principles for deformity correction to treat cubitus varus in children.

ELIGIBILITY:
Inclusion Criteria:

* surgery performed over 6 months after the occurrence of SHFs
* difference in flexion angles of the affected and unaffected limbs of >15 degrees
* recovery of elbow function pre-ostomy

Exclusion Criteria:

* any other surgical approach used
* consent not obtained from the patient's guardians
* incomplete follow-up

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All the patients were performed surgery between July 2015 and October 2017
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Elbow appearance | 3th month after surgery
  elbows were evaluated using radiography and appearence

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No